CLINICAL TRIAL: NCT00569244
Title: A Multi-center, Open-label, Randomized, Controlled, Parallel-group Study to Assess Efficacy and Safety of an Extended Flexible Regimen of the Combined Oral Contraceptive SH T00186D (0.02 mg Ethinylestradiol as Beta-cyclodextrin Clathrate and 3 mg Drospirenone) Compared to the Conventional Regimen of SH T00186D in the Treatment of Primary Dysmenorrhea
Brief Title: SH T00186 in the Treatment of Primary Dysmenorrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91587; 2006-004899-13 (EudraCT Number); 310882 (Other: Company Internal)
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Primary Dysmenorrhea
Keywords: Primary Dysmenorrhea; Menstrual Pain; Oral Contraception
MeSH Terms: conditions — Dysmenorrhea | interventions — drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Drug: YAZ flex (SH T00186D)
- Arm 2 (Active Comparator)
  Interventions: Drug: YAZ (SH T00186D)

INTERVENTIONS:
Drug: Drug: YAZ flex (SH T00186D) — Extended flexible regimen of YAZ (SH T00186D); triggered by bleeding events(Tablet p.o. (oral))
  Arms: Arm 1
Drug: YAZ (SH T00186D) — YAZ (SH T 00186D) administered in the conventional regimen (24 days active + 4 days placebo) (Tablet p.o. (oral))
  Arms: Arm 2

SUMMARY:
The investigational drug SH T00186D is an oral contraceptive. The investigational drug used in this study contains the estrogen ethinylestradiol (EE) and the progestogen drospirenone (DRSP).

The aim of the present study is to evaluate efficacy and safety of the investigational drug in the treatment of menstrual pain (pelvic pain occurring shortly before, at onset, during menstruation). Two different regimens of intake of the same investigational product will be compared.

Patients have to undergo 2 -3 Baseline cycles (depending on whether the patient was an OC user before), during which menstrual pain, bleeding events, and pain killer intake have to be documented. During this observation period, the intake of hormonal contraceptives is not allowed. Other contraceptive methods (condoms with spermicide, pessary with spermicide) have to be used. If the patient is eligible for the study, she will be randomly assigned to one of the two treatment groups. Treatment group A will take the medication according to an extended flexible regimen, i.e., tablet intake will be triggered by bleeding events. Treatment group B will take the study medication in the 24 + 4 days regimen. That means, tablets to be taken on cycle days 1 - 24 contain the hormone combination, whereas tablets 25 - 28 do not contain any active ingredients, i.e., these are so called placebo tablets.

Treatment will last at least 140 days, but can be prolonged in Treatment Group A depending of occurrence of menstrual bleeding. The overall study duration will be 10 months for each patient.

During the whole study period, 5 visits are planned. At Screening and Final examination, a thorough physical examination and a gynecological examination (including breath palpation and cervical smear ) will be performed. Blood samples will be taken for safety laboratory parameters.

Additional examinations can be performed any time, if this becomes necessary for medical reasons.

Patients will be provided with a patient diary to document the intake of study medication, any bleeding events and days without bleeding, pregnancy test results, any dysmenorrheic (menstrual) pain and its intensity and its interference with daily activity, and intake of pain medication. The pain medication (ibuprofen) will be provided.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy female patients with moderate to severe primary dysmenorrhea
* Prospective self-rated sum pain score of >/= 8 during the 2 baseline cycles
* Age between 18 and 40 years (inclusive) with smoking habits as follows:

  * between 18 and 30 years of age. daily cigarette consumption not above 10
  * above 30 years of age, no smoking

Exclusion Criteria:

* Current signs of history of any forms of secondary dysmenorrhea
* Any concomitant disease of condition that requires any intake of analgesic medication
* Occurrence of less than six menstrual cycles before Visit 1 following delivery, abortion, or lactation
* Clinically significant depression

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 223 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Number of days with dysmenorrheic pain | 140 days

SECONDARY OUTCOMES:
Use of rescue medication | 140 days
Interference with daily activity | 140 days
Number of days: with at least moderate dysmenorrheic pain | 140 days
Number of days with pelvic pain | 140 days
Number of days with dysmenorrheic pain associated with withdrawal bleeding | 140 days
Number of days with dysmenorrheic pain associated with unscheduled bleeding | 140 days
Bleeding patterns | Whole treatment period
Assessment of treatment | Whole treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (19):
- Germany (16):
  - Heidelberg, Baden-Wurttemberg
  - Nuremberg, Bavaria
  - Frankfurt am Main, Hesse
  - Fulda, Hesse
  - Mühlheim am Main, Hesse
  - Hanover, Lower Saxony
  - Leipzig, Saxony
  - Wurzen, Saxony
  - Bernburg, Saxony-Anhalt
  - Blankenburg, Saxony-Anhalt
  - Burg, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Gera, Thuringia
  - Kahla, Thuringia
- United Kingdom (3):
  - Chesterfield, Derbyshire
  - Newcastle upon Tyne, Tyne and Wear
  - London

REFERENCES:
- [Result] Strowitzki T, Kirsch B, Elliesen J. Efficacy of ethinylestradiol 20 mug/drospirenone 3 mg in a flexible extended regimen in women with moderate-to-severe primary dysmenorrhoea: an open-label, multicentre, randomised, controlled study. J Fam Plann Reprod Health Care. 2012 Apr;38(2):94-101. doi: 10.1136/jfprhc-2011-100225. PMID 22454006
- [Derived] Schroll JB, Black AY, Farquhar C, Chen I. Combined oral contraceptive pill for primary dysmenorrhoea. Cochrane Database Syst Rev. 2023 Jul 31;7(7):CD002120. doi: 10.1002/14651858.CD002120.pub4. PMID 37523477
- See also: Click here and search for information of Bayer products for Europe — http://www.clinicaltrialsregister.eu